CLINICAL TRIAL: NCT07295106
Title: Evaluation of the Effects of Personalized Music Therapy on Preterm Infants Admitted to the Neonatal Intensive Care Unit (NICU) and on Parental Stress: A Pilot Randomized Crossover Controlled Trial
Brief Title: Personalized Music Therapy for Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fabrizio Faina (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Sponsor-Investigator, Fabrizio Faina, Registered Nurse (RN), Azienda Ospedaliera di Perugia; Program Coordinator, Degree Program in Nursing, University of Perugia; Sponsor-Investigator, Azienda Ospedaliera di Perugia
Organization: Azienda Ospedaliera di Perugia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MTR20245CLO; CE-1558/24 (Other: Comitato Etico Regionale Umbria); CET-4855/24 (Other: Comitato Etico Regionale Umbria)
Record Dates: First submitted 2025-11-23; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Infant, Premature; Stress, Psychological
Keywords: Neonatal Intensive Care Unit; NICU; Music Therapy; Parental Voice; Tissue Oxygenation Index (TOI); Respiratory Rate; Near-Infrared Spectroscopy (NIRS); Heart Rate; Oxygen Saturation
MeSH Terms: conditions — Premature Birth; Stress, Psychological | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB: PMT then Quiet Rest (Experimental): Two period crossover. Period 1 = Personalized Music Therapy (PMT) during Phase 2 (10 to 40 min); Period 2 = Quiet Rest during Phase 2 (10 to 40 min). Washout between periods = 2 days. Each Period lasts 50 minutes (0 to 9 min Acclimation Rest; 10 to 40 min Treatment Exposure; 40 to 50 min Post-Exposure Rest). Measurements summarized as 5 minute window means at 5 to 9, 21 to 25, and 46 to 50 minutes.
  Interventions: Behavioral: Personalized Music Therapy (PMT); Behavioral: Quiet Rest
- Sequence BA: Quiet Rest then PMT (Experimental): Two period crossover. Period 1 = Quiet Rest during Phase 2 (10 to 40 min); Period 2 = Personalized Music Therapy (PMT) during Phase 2 (10 to 40 min). Washout between periods = 2 days. Each Period lasts 50 minutes (0 to 9 min Acclimation Rest; 10 to 40 min Treatment Exposure; 40 to 50 min Post-Exposure Rest). Measurements summarized as 5 minute window means at 5 to 9, 21 to 25, and 46 to 50 minutes.
  Interventions: Behavioral: Personalized Music Therapy (PMT); Behavioral: Quiet Rest

INTERVENTIONS:
Behavioral: Personalized Music Therapy (PMT) — Personalized Music Therapy (PMT): playback of the parent's recorded voice during Phase 2 (10 to 40 minutes) within a standardized 50 minute Period conducted in a low stimulation NICU room. Audio is prepared in advance by a trained music therapist (smoothing peaks, removing artifacts, setting a target level). Delivered via bedside speaker positioned approximately 30 cm from the infant's head; target intensity approximately 45 dBA (plus or minus 3 dB) at the infant's ear level. Phase 1 (0 to 9 minutes) and Phase 3 (40 to 50 minutes) are rest without added stimulation per protocol and are not part of the PMT exposure.
  Other Names: Music Therapy; Parental voice
Behavioral: Quiet Rest — Quiet Rest: low stimulation rest during Phase 2 (10 to 40 minutes) within the same standardized 50 minute Period used for PMT. Phase 1 (0 to 9 minutes) and Phase 3 (40 to 50 minutes) are also rest without added stimulation. Room conditions and handling minimization match those used for PMT.

SUMMARY:
Preterm infants in the Neonatal Intensive Care Unit (NICU) face environmental and clinical stressors that may affect physiological stability and development. This pilot randomized crossover study tests Personalized Music Therapy (PMT) based on recorded parental voices versus Quiet Rest. Outcomes include tissue oxygenation index (TOI) via near-infrared spectroscopy (NIRS) and heart rate (HR), respiratory rate (RR), and oxygen saturation (SpO2). Each infant completes two Periods (PMT and Quiet Rest) in randomized order, separated by a 2-day washout. Parental stress is measured at discharge using the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU). Findings inform feasibility, variance estimates, and protocol refinements for a larger trial.

DETAILED DESCRIPTION:
Background and rationale. Preterm infants in the Neonatal Intensive Care Unit (NICU) are exposed to noise, light, and frequent handling, which can affect physiology and development and increase parental distress. Family-centered music therapy using the parental voice is a low-risk intervention that may modulate cerebral oxygenation and autonomic parameters during exposure. Neonatal NIRS studies report small-to-moderate average changes in cerebral oxygenation with parental voice or music and heterogeneous individual responses, supporting standardized procedures and within-participant designs (van Bel 2008; Alderliesten 2016; Meder 2021; Yue 2021).

Ethics and consent. Enrollment proceeds under Ethics Committee approval on file; written informed consent is obtained from the parent(s) or legal guardian(s) per local policy. Consent from both parents is sought when applicable; a single signature is acceptable in single-parent or court-sanctioned guardianship cases according to site policy.

Design. Single-center, randomized 2 by 2 crossover pilot. Infants are randomized to Sequence AB (Period 1 = PMT, washout 2 days, Period 2 = Quiet Rest) or Sequence BA (Period 1 = Quiet Rest, washout 2 days, Period 2 = PMT).

Pre-intervention voice preparation (outside study periods). A trained music therapist records the parent's singing or voice and performs basic audio processing (smoothing peaks, removing artifacts, setting a target intensity). The audio files are stored securely for audio playback during PMT. No outcomes are collected during preparation.

Conduct of each period (50 minutes, 8:00 to 9:00 PM local time, low-stimulation NICU room). A bedside speaker is positioned approximately 30 cm from the infant's head; audio playback is set to approximately 45 dBA (plus or minus 3) at the infant's ear level. Each period follows the same structure:

* Phase 1 (0 to 9 minutes): Acclimation Rest (no stimulation)
* Phase 2 (10 to 40 minutes): Treatment Exposure (PMT or Quiet Rest, per randomized sequence)
* Phase 3 (40 to 50 minutes): Post-Exposure Rest (no stimulation) Measurements within each period. TOI (NIRS), HR, RR, and SpO2 are summarized as 5-minute window means at minutes 5 to 9 (Phase 1), minutes 21 to 25 (Phase 2), and minutes 46 to 50 (Phase 3). A 2-day washout separates periods to mitigate carryover.

Stopping criteria and resumption. Stop immediately if any of the following occurs: SpO2 below 85 percent for 30 seconds or more, or below 88 percent persistent; HR below 100 beats per minute for 30 seconds or more, or above 200 beats per minute persistent; apnea 20 seconds or longer, or RR 80 breaths per minute or higher persistent; cyanosis, marked pallor, hypotonia, or inconsolable irritability or crying; urgent procedures or non-deferrable handling; intolerance to the acoustic stimulus (for example, marked agitation or avoidance); parent request, if present. Resumption occurs only after clinical reassessment by the attending neonatologist or covering clinician and stabilization (parameters within safety ranges for 5 minutes or more). Nurses and physicians are authorized to stop according to criteria.

Parental stress. At discharge, parents complete the PSS:NICU as a self-report questionnaire assisted by trained NICU staff (for example, a nurse or psychologist).

Sample size. This 2 by 2 crossover pilot focuses on feasibility and estimation of the within-participant variance and effect magnitude on TOI. Based on NICU NIRS literature-small average changes in cerebral oxygenation with parental voice or music and non-trivial within-participant variability unless procedures are standardized-a clinically relevant within-participant mean difference (delta) of about 3 TOI percentage points (PMT minus Quiet Rest during minutes 21 to 25) and an expected within-participant standard deviation of approximately 4 to 5 points are assumed under standardized procedures (fixed time windows, low-stimulation room, consistent sensor placement, artifact rules). With 20 infants, the approximate 95 percent confidence-interval half-width is about 1.96 divided by the square root of 20 times the standard deviation (about 0.44 times SD), yielding roughly plus or minus 1.8 to 2.2 percentage points if SD is 4 to 5. This precision is acceptable for a pilot focused on estimation and feasibility and will inform sizing of a subsequent confirmatory trial (van Bel 2008; Alderliesten 2016; Meder 2021; Yue 2021).

Statistical analysis. The primary estimand is the within-participant mean difference (PMT minus Quiet Rest) in TOI during minutes 21 to 25 (5-minute window). The primary analysis uses a linear mixed-effects model with fixed effects for treatment (PMT versus Quiet Rest), period (1 versus 2), and sequence (AB versus BA), and a random intercept for participant. First-order carryover is assessed; if present, a sensitivity analysis restricted to Period 1 is reported. Secondary endpoints are exploratory and are analyzed analogously; multiplicity adjustments are not applied unless specified in the Statistical Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants admitted to the Neonatal Intensive Care Unit (NICU) of Azienda Ospedaliera di Perugia, Santa Maria della Misericordia, Perugia (Italy) at the time of enrollment.
* Gestational age at birth 28+0 to 36+6 weeks.
* Age at enrollment: 5 to 15 days.
* Stable vital signs at enrollment per unit policy.
* Apgar score at 5 minutes ≥ 7.
* Birth weight appropriate for gestational age, between the 50th and 90th percentile.
* Written informed consent from parent(s) or legal guardian(s).

Exclusion Criteria:

* Post-operative status at the time of enrollment.
* One or more of the following: intraventricular hemorrhage, necrotizing enterocolitis, sepsis, significant pulmonary disease, or neonatal anemia.
* Congenital anomalies.
* Hypersensitivity or intolerance to sound.
* Maternal history of drug and/or alcohol misuse during pregnancy.
* Lack of parental consent.

Ages: 5 Days to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
TOI 21 to 25 min | Minutes 21-25 of each 50-minute Period (Phase 2)
  Mean tissue oxygenation index (TOI, percent) over minutes 21 to 25. Primary comparison is the within-participant difference (PMT minus Quiet Rest) in a two-sequence, two-period crossover.

SECONDARY OUTCOMES:
TOI 5 to 9 min | Minutes 5-9 of each 50-minute Period (Phase 1)
  Mean tissue oxygenation index (TOI, percent) over minutes 5 to 9. Within-participant difference (PMT minus Quiet Rest).
TOI 46 to 50 min | Minutes 46-50 of each 50-minute Period (Phase 3)
  Mean tissue oxygenation index (TOI, percent) over minutes 46 to 50. Within-participant difference (PMT minus Quiet Rest).
HR 5 to 9 min | Minutes 5-9 of each 50-minute Period (Phase 1)
  Mean heart rate (HR, beats per minute) over minutes 5 to 9. Within-participant difference (PMT minus Quiet Rest).
HR 21 to 25 min | Minutes 21-25 of each 50-minute Period (Phase 2)
  Mean heart rate (HR, beats per minute) over minutes 21 to 25. Within-participant difference (PMT minus Quiet Rest).
HR 46 to 50 min | Minutes 46-50 of each 50-minute Period (Phase 3)
  Mean heart rate (HR, beats per minute) over minutes 46 to 50. Within-participant difference (PMT minus Quiet Rest).
RR 5 to 9 min | Minutes 5 to 9 of each 50-minute Period (Phase 1)
  Mean respiratory rate (RR, breaths per minute) over minutes 5 to 9. Within-participant difference (PMT minus Quiet Rest).
RR 21 to 25 min | Minutes 21-25 of each 50-minute Period (Phase 2)
  Mean respiratory rate (RR, breaths per minute) over minutes 21 to 25. Within-participant difference (PMT minus Quiet Rest).
RR 46 to 50 min | Minutes 46-50 of each 50-minute Period (Phase 3)
  Mean respiratory rate (RR, breaths per minute) over minutes 46 to 50. Within-participant difference (PMT minus Quiet Rest).
SpO2 5 to 9 min | Minutes 5 to 9 of each 50-minute Period (Phase 1)
  Mean oxygen saturation (SpO2, percent) over minutes 5 to 9. Within-participant difference (PMT minus Quiet Rest).
SpO2 21 to 25 min | Minutes 21 to 25 of each 50-minute Period (Phase 2)
  Mean oxygen saturation (SpO2, percent) over minutes 21 to 25. Within-participant difference (PMT minus Quiet Rest).
SpO2 46 to 50 min | Minutes 46-50 of each 50-minute Period (Phase 3)
  Mean oxygen saturation (SpO2, percent) over minutes 46 to 50. Within-participant difference (PMT minus Quiet Rest).
PSS:NICU | Immediately after the intervention
  Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) total score; higher scores indicate greater perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Unit (NICU), Ospedale Santa Maria della Misericordia - Azienda Ospedaliera di Perugia, Perugia, PG, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared because this study involves a small and vulnerable population (preterm infants), and full de-identification cannot be ensured.

REFERENCES:
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Yue W, Han X, Luo J, Zeng Z, Yang M. Effect of music therapy on preterm infants in neonatal intensive care unit: Systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2021 Feb;77(2):635-652. doi: 10.1111/jan.14630. Epub 2020 Nov 17. PMID 33200833
- [Background] Alderliesten T, Dix L, Baerts W, Caicedo A, van Huffel S, Naulaers G, Groenendaal F, van Bel F, Lemmers P. Reference values of regional cerebral oxygen saturation during the first 3 days of life in preterm neonates. Pediatr Res. 2016 Jan;79(1-1):55-64. doi: 10.1038/pr.2015.186. Epub 2015 Sep 21. PMID 26389823
- [Background] van Bel F, Lemmers P, Naulaers G. Monitoring neonatal regional cerebral oxygen saturation in clinical practice: value and pitfalls. Neonatology. 2008;94(4):237-44. doi: 10.1159/000151642. Epub 2008 Sep 11. PMID 18784420
- [Background] Meder U, Tarjanyi E, Kovacs K, Szakmar E, Cseko AJ, Hazay T, Belteki G, Szabo M, Jermendy A. Cerebral oxygenation in preterm infants during maternal singing combined with skin-to-skin care. Pediatr Res. 2021 Oct;90(4):809-814. doi: 10.1038/s41390-020-01235-2. Epub 2020 Dec 1. PMID 33262445